CLINICAL TRIAL: NCT06279416
Title: Evaluation of Advanced Airway Methods Applied to Patients Who Were Awakened Due to Difficult Airway in Another Center or Who Were Predicted to Have Difficult Airway in Preoperative Evaluation
Brief Title: Expected Difficult Airway Management
Status: Completed | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-31
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Awake Intubation; Advanced Airway Techniques
Keywords: videolaryngoscopy; fiberoptic bronchoscope; supraglottic airway device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- grup-1: awake nasal fiberoptic intubation: awake nasal fiberoptic intubation
  Interventions: Procedure: fiberoptic intubation
- grup-2: awake intubation with laryngeal mask airway-mediated aintree catheter: awake intubation with laryngeal mask airway-mediated aintree catheter
  Interventions: Procedure: laryngeal mask airway-mediated aintree catheter
- grup-3: awake intubation with videolaryngoscopy: awake intubation with videolaryngoscopy
  Interventions: Procedure: videolaryngoscopy

INTERVENTIONS:
Procedure: fiberoptic intubation — awake nasal fiberoptic intubation
  Groups: grup-1: awake nasal fiberoptic intubation
Procedure: laryngeal mask airway-mediated aintree catheter — awake intubation with laryngeal mask airway-mediated aintree catheter
  Groups: grup-2: awake intubation with laryngeal mask airway-mediated aintree catheter
Procedure: videolaryngoscopy — awake intubation with videolaryngoscopy
  Groups: grup-3: awake intubation with videolaryngoscopy

SUMMARY:
In this study, the investigators will evaluate the advanced airway methods applied in the anesthesiology and reanimation clinic of the hospital to patients who met the criteria for awake intubation specified in the ASA 2022 difficult airway management guideline or who could not be intubated after induction of anesthesia in another center. The advanced airway method applied to the difficult airway patient expected in the operating room, the duration, success and complications of the method will be observed and recorded.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be informed about the difficult airway and their verbal and written consent will be obtained.

When participants are taken to the room, an observer will be in the operation room. There was no emergency to the patient's primary anesthesiologist, will not be involved. Record patients' demographic data, Mallampati scores, thyromental distance, and neck circumference.

The airway method preferred by the physician, procedure duration, number of attempts, success, and complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Meets the expected difficult airway criteria
* Being awakened after induction of anesthesia in another center
* At least one of the awake intubation criteria in the DAS 2022 guideline
* Elective surgeries

Exclusion Criteria:

* Emergency surgeries
* Patients intubated with anesthesia
* Noncoopere patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were previously evaluated for difficult airway criteria and predicted to have a difficult airway or who could not be ventilated or intubated after induction of anesthesia in another center.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of advanced airway methods in the awake patient with difficult airway. | 1 year
  Comparison of the superiority of advanced airway methods applied to the expected difficult airway patient in the operating room. The number of attempts and duration for successful intubation between groups will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yilmaz, Principal Investigator — Kocaeli City Hospital Anesthesiology and Reanimation
Locations (1):
- Kocaeli City Hospital, Kocaeli, Turkey (Türkiye)